CLINICAL TRIAL: NCT05478707
Title: Therapeutic Strategies for Microvascular Dysfunction in Type 1 Diabetes
Acronym: KML002
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Institution transfer
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kaitlin Love, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 210198
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1; Endothelial Dysfunction
Keywords: microvessels; oxidative stress; Dulaglutide; Glucagon-like peptide-1; Exercise therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants randomized to dulaglutide or placebo and study personnel who analyze data and instruct patients regarding insulin adjustments will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Saline subcutaneous injection, volume matched to dulaglutide, i.e. 0.5 mL weekly for 14 weeks
  Interventions: Drug: Placebo
- Dulaglutide (Active Comparator): Dulaglutide (0.75 mg/0.5 mL weekly for 2 weeks, then 1.5 mg/0.5 mL weekly for 12 weeks) subcutaneous injection
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Dulaglutide — GLP1-RA
  Arms: Dulaglutide
Drug: Placebo — Saline placebo
  Arms: Placebo

SUMMARY:
The investigators will test the hypothesis that, in adults with type 1 diabetes (T1D), glucagon-like peptide-1 receptor agonism (GLP-1RA, i.e. dulaglutide) enhances insulin-mediated skeletal muscle microvascular perfusion via attenuating endothelial oxidative stress and thereby improving endothelial function.

DETAILED DESCRIPTION:
In this study, 47 (n=32 needed to complete) adult participants with type 1 diabetes will be randomized (1:1) to 14-weeks of one of 2 interventions: 1) dulaglutide, 2) placebo.

Participants will undergo two study admissions at baseline and 14 weeks. Prior to each admission, participants will wear a continuous glucose monitor (Dexcom G6 Professional) for 10 days to assess glycemic variability (GV). Prior to admissions, they will undergo cardiorespiratory fitness testing. On study admission days, participants will undergo an antecubital vein endothelial cell biopsy prior to commencing vascular testing. From the harvested endothelial cells, the investigators will quantify endothelial cell reactive oxygen species (ROS) and gene expression relevant to insulin-mediated endothelial function. Vascular testing will include contrast enhanced ultrasound of quadriceps muscle to determine microvascular blood volume (MBV). The investigators will also measure brachial artery flow mediated dilation (FMD). Quadriceps skeletal muscle oxygenation (HHb) will also be measured. These vascular and muscle oxygenation measurements will be conducted before and after a 120-minute euglycemic insulin clamp which will measure insulin sensitivity based on glucose infusion rate (GIR).

This randomized, placebo-controlled study will assess whether GLP-1 receptor agonism with dulaglutide or exercise training improves insulin-mediated skeletal muscle microvascular perfusion. The investigators will assess for predictive relationships between microvascular perfusion and cardiorespiratory fitness (VO2max), insulin sensitivity (GIR), endothelial reactive oxygen species (ROS), and glycemic variability (GV).

ELIGIBILITY:
Inclusion criteria:

* History of type 1 diabetes, duration > 5 years
* Age 18-40 years
* HbA1c < 8.5%
* BMI 19-34.9 kg/m2
* Using insulin for diabetes treatment only (multiple daily injections or insulin pump with or without sensor augmentation)
* On stable regimen of non-diabetic medications for the last 6 months
* All screening labs within normal limits or not clinically significant
* C-peptide <0.6 ng/ml

Exclusion criteria:

* Pregnancy or currently breastfeeding
* Smoking history within 6 months
* History of microvascular (microalbuminuria, retinopathy, neuropathy) or macrovascular diabetes complications (coronary artery disease, stroke, peripheral vascular disease) as well as clinically significant cardiac arrhythmias or conduction disorders
* Taking vasoactive medications (i.e. calcium channel blockers, angiotensin-converting enzyme or renin inhibitors, angiotensin-receptor blockers, nitrates, alpha-blockers).
* Known hypersensitivity to perflutren (contained in Definity© contrast)
* Screening O2 saturation <90%
* Musculoskeletal condition preventing participation in exercise testing or exercise training
* Acute or unstable disease other than T1D
* Hypoglycemia unawareness (based on Clarke's questionnaire)
* History of gastroparesis, severe gastroesophageal reflux, pancreatitis, personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2
* Anemia (hemoglobin <12 g/dL in women, hemoglobin <13 g/dL in men), eosinophilia (absolute eosinophil count >500 cells/microliter) leukopenia (total white blood cells <4,000 cells/microliter)
* Diabetic ketoacidosis (DKA) on presentation to screening visits or study admission days
* Hospital admission for DKA within 1 year

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular blood volume (MBV) | At baseline and after 14 weeks of treatment.
  Insulin mediated change in muscle microvascular blood volume (MBV). A measure of microvascular nitric oxide dependent endothelial function

SECONDARY OUTCOMES:
Brachial artery flow mediated dilation (FMD) | At baseline and after 14 weeks of treatment
  Post-occlusive percent (%) change in diameter. A measure of conduit artery nitric oxide-dependent endothelial function.
Glucose infusion rate (GIR) | At baseline and after 14 weeks of treatment
  Mean GIR over the final 30 minutes of euglycemic insulin clamp; a measure of insulin sensitivity
Cardiorespiratory fitness, maximum consumption of oxygen (VO2max) | At baseline and after 14 weeks of treatment
  Assessed by cycle ergometer exercise testing.
Skeletal muscle oxygenation, deoxyhemoglobin (HHb) | At baseline and after 14 weeks of treatment. Measured before and after insulin clamp.
  Assessed by frequency domain multi-distance near-infrared spectroscopy (NIRS) monitor at the quadriceps muscle

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlin Love, MD, Principal Investigator — Associate Professor - Endocrinology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Shinkai T, Saijo N, Tominaga K, Eguchi K, Shimizu E, Sasaki Y, Fujita J, Futami H. Comparison of vindesine plus cisplatin or vindesine plus mitomycin in the treatment of advanced non-small cell lung cancer. Cancer Treat Rep. 1985 Sep;69(9):945-51. PMID 2992785
- [Background] Harrison RM. Tissue-air ratios and scatter-air ratios for diagnostic radiology (1-4 mm Al HVL). Phys Med Biol. 1983 Jan;28(1):1-18. doi: 10.1088/0031-9155/28/1/001. PMID 6828554
- [Background] Furuyama F. Strain difference in thermoregulation of rats surviving extreme heat. J Appl Physiol Respir Environ Exerc Physiol. 1982 Feb;52(2):410-5. doi: 10.1152/jappl.1982.52.2.410. PMID 7061293
- [Background] Tabayashi K, McKeown PP, Miyamoto M, Luedtke AE, Thomas R, Allen MD, Misbach GA, Ivey TD. Ischemic myocardial protection. Comparison of nonoxygenated crystalloid, oxygenated crystalloid, and oxygenated fluorocarbon cardioplegic solutions. J Thorac Cardiovasc Surg. 1988 Feb;95(2):239-46. PMID 3339891
- [Background] Donga E, Dekkers OM, Corssmit EP, Romijn JA. Insulin resistance in patients with type 1 diabetes assessed by glucose clamp studies: systematic review and meta-analysis. Eur J Endocrinol. 2015 Jul;173(1):101-9. doi: 10.1530/EJE-14-0911. Epub 2015 Apr 21. PMID 25899581
- [Background] Kuijpers PJ, Lacquet LK, Skotnicki SH, Linssen GH, Vonk JT. Surgical treatment for acute myocardial ischaemia. J Cardiovasc Surg (Torino). 1974 Mar;15(2):209-10. No abstract available. PMID 4834265
- [Background] Xu TH, Xie DZ, Wan TB, Pai B, Wang LX. Studies on immunological changes among schizophrenic patients. Schizophr Res. 1988 Nov-Dec;1(6):431-3. doi: 10.1016/0920-9964(88)90026-6. No abstract available. PMID 3154531
- [Background] Poldermans D, Arnese M, Fioretti PM, Salustri A, Boersma E, Thomson IR, Roelandt JR, van Urk H. Improved cardiac risk stratification in major vascular surgery with dobutamine-atropine stress echocardiography. J Am Coll Cardiol. 1995 Sep;26(3):648-53. doi: 10.1016/0735-1097(95)00240-5. PMID 7642854
- [Background] Ce GV, Rohde LE, da Silva AM, Punales MK, de Castro AC, Bertoluci MC. Endothelial dysfunction is related to poor glycemic control in adolescents with type 1 diabetes under 5 years of disease: evidence of metabolic memory. J Clin Endocrinol Metab. 2011 May;96(5):1493-9. doi: 10.1210/jc.2010-2363. Epub 2011 Feb 23. PMID 21346068
- [Background] Inaba Y, Chen JA, Bergmann SR. Prediction of future cardiovascular outcomes by flow-mediated vasodilatation of brachial artery: a meta-analysis. Int J Cardiovasc Imaging. 2010 Aug;26(6):631-40. doi: 10.1007/s10554-010-9616-1. Epub 2010 Mar 26. PMID 20339920
- [Background] Mischler TW, Rubio B, Larranaga A, Guiloff E, Moggia AV. Further experience with quingestanol acetate as a postcoital oral contraceptive. Contraception. 1974 Mar;9(3):221-5. doi: 10.1016/0010-7824(74)90013-4. PMID 4613534
- [Background] Love KM, Jahn LA, Hartline LM, Patrie JT, Barrett EJ, Liu Z. Insulin-mediated muscle microvascular perfusion and its phenotypic predictors in humans. Sci Rep. 2021 Jun 1;11(1):11433. doi: 10.1038/s41598-021-90935-8. PMID 34075130
- [Background] Bertelli A, Giovannini L, Romano MR, Maltinti G, Dell'Osso L, Bertelli AA. Experimental comparative renal toxicity of lithium and rubidium. Drugs Exp Clin Res. 1985;11(4):269-73. PMID 3836129
- [Background] Akber SF. The physics of NMR tomography. Nuklearmedizin. 1986 Feb;25(1):33-8. PMID 3714509
- [Background] Saffari B, Jones LA, el-Naggar A, Felix JC, George J, Press MF. Amplification and overexpression of HER-2/neu (c-erbB2) in endometrial cancers: correlation with overall survival. Cancer Res. 1995 Dec 1;55(23):5693-8. PMID 7585656
- [Background] Liu HY, Cao SY, Hong T, Han J, Liu Z, Cao W. Insulin is a stronger inducer of insulin resistance than hyperglycemia in mice with type 1 diabetes mellitus (T1DM). J Biol Chem. 2009 Oct 2;284(40):27090-100. doi: 10.1074/jbc.M109.016675. Epub 2009 Aug 4. PMID 19654321
- [Background] Wang N, Tan AWK, Jahn LA, Hartline L, Patrie JT, Lin S, Barrett EJ, Aylor KW, Liu Z. Vasodilatory Actions of Glucagon-Like Peptide 1 Are Preserved in Skeletal and Cardiac Muscle Microvasculature but Not in Conduit Artery in Obese Humans With Vascular Insulin Resistance. Diabetes Care. 2020 Mar;43(3):634-642. doi: 10.2337/dc19-1465. Epub 2019 Dec 30. PMID 31888883
- [Background] Batchuluun B, Inoguchi T, Sonoda N, Sasaki S, Inoue T, Fujimura Y, Miura D, Takayanagi R. Metformin and liraglutide ameliorate high glucose-induced oxidative stress via inhibition of PKC-NAD(P)H oxidase pathway in human aortic endothelial cells. Atherosclerosis. 2014 Jan;232(1):156-64. doi: 10.1016/j.atherosclerosis.2013.10.025. Epub 2013 Nov 5. PMID 24401231
- [Background] Subaran SC, Sauder MA, Chai W, Jahn LA, Fowler DE, Aylor KW, Basu A, Liu Z. GLP-1 at physiological concentrations recruits skeletal and cardiac muscle microvasculature in healthy humans. Clin Sci (Lond). 2014 Aug;127(3):163-70. doi: 10.1042/CS20130708. PMID 24552454
- [Background] Lepore JJ, Olson E, Demopoulos L, Haws T, Fang Z, Barbour AM, Fossler M, Davila-Roman VG, Russell SD, Gropler RJ. Effects of the Novel Long-Acting GLP-1 Agonist, Albiglutide, on Cardiac Function, Cardiac Metabolism, and Exercise Capacity in Patients With Chronic Heart Failure and Reduced Ejection Fraction. JACC Heart Fail. 2016 Jul;4(7):559-566. doi: 10.1016/j.jchf.2016.01.008. Epub 2016 Mar 30. PMID 27039125
- [Background] Basu A, Charkoudian N, Schrage W, Rizza RA, Basu R, Joyner MJ. Beneficial effects of GLP-1 on endothelial function in humans: dampening by glyburide but not by glimepiride. Am J Physiol Endocrinol Metab. 2007 Nov;293(5):E1289-95. doi: 10.1152/ajpendo.00373.2007. Epub 2007 Aug 21. PMID 17711996
- [Background] Budalica M, Plamenac P, Tvrtkovic R, Gmaz-Nikulin E. [Cystic mediastinal lymphangioma]. Srp Arh Celok Lek. 1971 Jun;99(6):395-401. No abstract available. Serbian. PMID 5142002
- [Background] [Hazards to the conception product of drugs administered to the pregnant woman. I. Round table discussion]. Bull Fed Soc Gynecol Obstet Lang Fr. 1968;20(5):Suppl:288-95. No abstract available. French. PMID 5759220
- [Background] Irace C, De Luca S, Shehaj E, Carallo C, Loprete A, Scavelli F, Gnasso A. Exenatide improves endothelial function assessed by flow mediated dilation technique in subjects with type 2 diabetes: results from an observational research. Diab Vasc Dis Res. 2013 Jan;10(1):72-7. doi: 10.1177/1479164112449562. Epub 2012 Jun 25. PMID 22732108
- [Background] Kiraly JF, Becker CE, Williams HE. Diabetic ketoacidosis. A review of cases at a university medical center. Calif Med. 1970 Apr;112(4):1-9. PMID 4985288
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Hernandez AF, Green JB, Janmohamed S, D'Agostino RB Sr, Granger CB, Jones NP, Leiter LA, Rosenberg AE, Sigmon KN, Somerville MC, Thorpe KM, McMurray JJV, Del Prato S; Harmony Outcomes committees and investigators. Albiglutide and cardiovascular outcomes in patients with type 2 diabetes and cardiovascular disease (Harmony Outcomes): a double-blind, randomised placebo-controlled trial. Lancet. 2018 Oct 27;392(10157):1519-1529. doi: 10.1016/S0140-6736(18)32261-X. Epub 2018 Oct 2. PMID 30291013
- [Background] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Background] Gutniak M, Orskov C, Holst JJ, Ahren B, Efendic S. Antidiabetogenic effect of glucagon-like peptide-1 (7-36)amide in normal subjects and patients with diabetes mellitus. N Engl J Med. 1992 May 14;326(20):1316-22. doi: 10.1056/NEJM199205143262003. PMID 1348845
- [Background] Mochon MC, Leyva JA. A new spectrophotometric method for determining triglycerides in serum. Clin Chim Acta. 1984 Sep 29;142(2):281-5. doi: 10.1016/0009-8981(84)90387-5. No abstract available. PMID 6499209
- [Background] Farinha JB, Ramis TR, Vieira AF, Macedo RCO, Rodrigues-Krause J, Boeno FP, Schroeder HT, Muller CH, Boff W, Krause M, De Bittencourt PIH Jr, Reischak-Oliveira A. Glycemic, inflammatory and oxidative stress responses to different high-intensity training protocols in type 1 diabetes: A randomized clinical trial. J Diabetes Complications. 2018 Dec;32(12):1124-1132. doi: 10.1016/j.jdiacomp.2018.09.008. Epub 2018 Sep 19. PMID 30270019
- [Background] Tielemans SM, Soedamah-Muthu SS, De Neve M, Toeller M, Chaturvedi N, Fuller JH, Stamatakis E. Association of physical activity with all-cause mortality and incident and prevalent cardiovascular disease among patients with type 1 diabetes: the EURODIAB Prospective Complications Study. Diabetologia. 2013 Jan;56(1):82-91. doi: 10.1007/s00125-012-2743-6. Epub 2012 Oct 10. PMID 23052062
- [Background] Tikkanen-Dolenc H, Waden J, Forsblom C, Harjutsalo V, Thorn LM, Saraheimo M, Elonen N, Tikkanen HO, Groop PH; FinnDiane Study Group. Physical Activity Reduces Risk of Premature Mortality in Patients With Type 1 Diabetes With and Without Kidney Disease. Diabetes Care. 2017 Dec;40(12):1727-1732. doi: 10.2337/dc17-0615. Epub 2017 Oct 16. PMID 29038314
- [Background] Komatsu WR, Gabbay MA, Castro ML, Saraiva GL, Chacra AR, de Barros Neto TL, Dib SA. Aerobic exercise capacity in normal adolescents and those with type 1 diabetes mellitus. Pediatr Diabetes. 2005 Sep;6(3):145-9. doi: 10.1111/j.1399-543X.2005.00120.x. PMID 16109070
- [Background] Lespagnol E, Tagougui S, Fernandez BO, Zerimech F, Matran R, Maboudou P, Berthoin S, Descat A, Kim I, Pawlak-Chaouch M, Boissiere J, Boulanger E, Feelisch M, Fontaine P, Heyman E. Circulating biomarkers of nitric oxide bioactivity and impaired muscle vasoreactivity to exercise in adults with uncomplicated type 1 diabetes. Diabetologia. 2021 Feb;64(2):325-338. doi: 10.1007/s00125-020-05329-8. Epub 2020 Nov 21. PMID 33219433
- [Background] Turinese I, Marinelli P, Bonini M, Rossetti M, Statuto G, Filardi T, Paris A, Lenzi A, Morano S, Palange P. "Metabolic and cardiovascular response to exercise in patients with type 1 diabetes". J Endocrinol Invest. 2017 Sep;40(9):999-1005. doi: 10.1007/s40618-017-0670-6. Epub 2017 Apr 6. PMID 28386795
- [Background] Eckstein ML, Farinha JB, McCarthy O, West DJ, Yardley JE, Bally L, Zueger T, Stettler C, Boff W, Reischak-Oliveira A, Riddell MC, Zaharieva DP, Pieber TR, Muller A, Birnbaumer P, Aziz F, Brugnara L, Haahr H, Zijlstra E, Heise T, Sourij H, Roden M, Hofmann P, Bracken RM, Pesta D, Moser O. Differences in Physiological Responses to Cardiopulmonary Exercise Testing in Adults With and Without Type 1 Diabetes: A Pooled Analysis. Diabetes Care. 2021 Jan;44(1):240-247. doi: 10.2337/dc20-1496. Epub 2020 Nov 12. PMID 33184152
- [Background] Olsen PR, Iversen HG, Hansen RI, Wolf H. [A simple preoperative ultrasonic method of estimating the size of the prostate]. Ugeskr Laeger. 1984 Dec 10;146(50):3899-901. No abstract available. Danish. PMID 6084353
- [Background] Schmidtke JR, Dixon FJ. The functional capacity of x-irradiated macrophages. J Immunol. 1972 Jun;108(6):1624-30. No abstract available. PMID 4113177
- [Background] Archer-Duste H. Clinical ethics: a mandate for nursing. J Perinat Neonatal Nurs. 1988 Jan;1(3):49-56. doi: 10.1097/00005237-198801000-00007. No abstract available. PMID 3379600
- [Background] Wei K, Jayaweera AR, Firoozan S, Linka A, Skyba DM, Kaul S. Quantification of myocardial blood flow with ultrasound-induced destruction of microbubbles administered as a constant venous infusion. Circulation. 1998 Feb 10;97(5):473-83. doi: 10.1161/01.cir.97.5.473. PMID 9490243
- [Background] Vincent MA, Clerk LH, Lindner JR, Klibanov AL, Clark MG, Rattigan S, Barrett EJ. Microvascular recruitment is an early insulin effect that regulates skeletal muscle glucose uptake in vivo. Diabetes. 2004 Jun;53(6):1418-23. doi: 10.2337/diabetes.53.6.1418. PMID 15161743
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Greenberg RN, Reilly PM, Weinandt WJ, Wilson KM, Bollinger M, Ojile JM. Comparison trial of clindamycin with aztreonam or gentamicin in the treatment of postpartum endometritis. Clin Ther. 1987;10(1):36-9. PMID 3329963
- [Background] Specter SC, Klein TW, Newton C, Mondragon M, Widen R, Friedman H. Marijuana effects on immunity: suppression of human natural killer cell activity of delta-9-tetrahydrocannabinol. Int J Immunopharmacol. 1986;8(7):741-5. doi: 10.1016/0192-0561(86)90010-x. PMID 3023245
- [Background] Herranz Jordan B, Bermudez-Canete Fernandez R, Herraiz Sarachaga JI, Acerete Guillen F, Bialkowski J, Gonzalez Dieguez C, Sanchez Fernandez PA, Diez Balda JI, Quero Jimenez M. [Non-surgical extraction of intravascular foreign bodies in children. Experience with 8 cases]. Rev Esp Cardiol. 1995 May;48(5):326-32. Spanish. PMID 7792427
- [Background] Crisci I, Aragona M, Politi KS, Daniele G, Del Prato S. GLP-1 receptor agonists in type 1 diabetes: a proof-of-concept approach. Acta Diabetol. 2015 Dec;52(6):1129-33. doi: 10.1007/s00592-015-0800-6. Epub 2015 Aug 21. PMID 26293127
- [Background] Mathieu C, Zinman B, Hemmingsson JU, Woo V, Colman P, Christiansen E, Linder M, Bode B; ADJUNCT ONE Investigators. Efficacy and Safety of Liraglutide Added to Insulin Treatment in Type 1 Diabetes: The ADJUNCT ONE Treat-To-Target Randomized Trial. Diabetes Care. 2016 Oct;39(10):1702-10. doi: 10.2337/dc16-0691. Epub 2016 Aug 9. PMID 27506222
- [Background] Ahren B, Hirsch IB, Pieber TR, Mathieu C, Gomez-Peralta F, Hansen TK, Philotheou A, Birch S, Christiansen E, Jensen TJ, Buse JB; ADJUNCT TWO Investigators. Efficacy and Safety of Liraglutide Added to Capped Insulin Treatment in Subjects With Type 1 Diabetes: The ADJUNCT TWO Randomized Trial. Diabetes Care. 2016 Oct;39(10):1693-701. doi: 10.2337/dc16-0690. Epub 2016 Aug 4. PMID 27493132
- [Background] Scott SN, Cocks M, Andrews RC, Narendran P, Purewal TS, Cuthbertson DJ, Wagenmakers AJM, Shepherd SO. High-Intensity Interval Training Improves Aerobic Capacity Without a Detrimental Decline in Blood Glucose in People With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Feb 1;104(2):604-612. doi: 10.1210/jc.2018-01309. PMID 30281094
- [Background] Lim F, Yang CZ, Cooper SL. Synthesis, characterization and ex vivo evaluation of polydimethylsiloxane polyurea-urethanes. Biomaterials. 1994 May;15(6):408-16. doi: 10.1016/0142-9612(94)90218-6. PMID 8080930
- [Background] Easty GC, Easty DM, Tchao R. The growth of heterologous tumour cells in chick embryos. Eur J Cancer (1965). 1969 Jun;5(3):287-95. doi: 10.1016/0014-2964(69)90079-6. No abstract available. PMID 5786070
- [Background] Jordan EM, Breen GA. Upstream region of a nuclear gene encoding the alpha-subunit of the human mitochondrial F0F1 ATP synthase. Biochim Biophys Acta. 1993 Apr 29;1173(1):115-7. doi: 10.1016/0167-4781(93)90256-d. PMID 8387339
- [Background] Travers GR, Ammon RG. The sodium hydroxide chemical matricectomy procedure. J Am Podiatry Assoc. 1980 Sep;70(9):476-8. doi: 10.7547/87507315-70-9-476. No abstract available. PMID 7440891
- [Background] Bally L, Zueger T, Buehler T, Dokumaci AS, Speck C, Pasi N, Ciller C, Paganini D, Feller K, Loher H, Rosset R, Wilhelm M, Tappy L, Boesch C, Stettler C. Metabolic and hormonal response to intermittent high-intensity and continuous moderate intensity exercise in individuals with type 1 diabetes: a randomised crossover study. Diabetologia. 2016 Apr;59(4):776-84. doi: 10.1007/s00125-015-3854-7. Epub 2016 Jan 6. PMID 26739816
- [Background] Martins EM, dos Santos RR, Moraes WB. [Biochemical aspects of resistance mechamism of mango (mangifera indica l. to ceratocystis fimbriata ell. & hals]. Arq Inst Biol (Sao Paulo). 1974 Oct-Dec;41(4):175-83. No abstract available. Portuguese. PMID 4461018
- [Background] Colombo PC, Ashton AW, Celaj S, Talreja A, Banchs JE, Dubois NB, Marinaccio M, Malla S, Lachmann J, Ware JA, Le Jemtel TH. Biopsy coupled to quantitative immunofluorescence: a new method to study the human vascular endothelium. J Appl Physiol (1985). 2002 Mar;92(3):1331-8. doi: 10.1152/japplphysiol.00680.2001. PMID 11842075
- [Background] Fox E, Abbatte EA, Said-Salah, Constantine NT, Wassef HH, Woody JN. Viral hepatitis markers in Djibouti: an epidemiological survey. Trans R Soc Trop Med Hyg. 1988;82(5):750-2. doi: 10.1016/0035-9203(88)90225-8. PMID 2855282